CLINICAL TRIAL: NCT06392581
Title: Prospective Observational Study on the Incidence of Invasive Fungal Infections in Patients With Ph-negative Acute Lymphoblastic Leukemia
Brief Title: Observational Study on Invasive Fungal Infection Incidence in Ph-neg Acute Lymphoblastic Leukemia Patients
Acronym: ALL-IFI
Status: Recruiting | Type: Observational
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Chiara Cattaneo, Head of Hematology inpatient unit, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: SEIFEM ALL-IFI 2022_NP 5250
Record Dates: First submitted 2024-03-01; First posted 2024-04-30 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Acute Lymphoblastic Leukemia
Keywords: invasive fungal infections; acute lymphoblastic leukemia; outcome
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Primary objective To document the occurrence of fungal infections during the early stages of chemotherapy (from onset to TP2, i.e., week 16) in adult Ph-neg ALL patients Secondary objectives

* To document the occurrence of IFI in relation to antifungal prophylaxis adopted
* To document the occurrence of IFI in relation to the age of the patients
* Document the occurrence of IFI in relation to the duration of neutropenia
* Document the occurrence of IFI in relation to the type of steroid treatment adopted (dexamethasone yes vs no)
* Document any delays in the initiation of consolidation chemotherapy in LLA patients with IFI
* Document the outcome of patients with ALL with IFI

Study design The study is prospective and observational, multicenter, real-life study involving 26 centers afferent to the SEIFEM group. All Ph-neg ALL patients aged 18 years or older treated with intensive chemotherapy starting from 01.06.22 for the duration of 18 months (+12 months follow-up) will be enrolled. The diagnosis of IFI will be defined according to EORTC 2019 criteria. Clinical information will be collected in paper CRFs, compiled anonymously.

The incidence of IFI and pulmonary aspergillosis during induction chemotherapy will be related to the following variables:

* Age
* Sex
* Type of AF prophylaxis performed
* LLA risk classification according to ESMO 2016 criteria
* Dose of dexamethasone administered
* Duration of neutropenia
* Hematologic and molecular response

DETAILED DESCRIPTION:
Primary objective To document the occurrence of fungal infections during the early stages of chemotherapy (from onset to TP2, i.e., week 16) in adult Ph-neg ALL patients Secondary objectives

* To document the occurrence of IFI in relation to antifungal prophylaxis adopted
* To document the occurrence of IFI in relation to the age of the patients
* Document the occurrence of IFI in relation to the duration of neutropenia
* Document the occurrence of IFI in relation to the type of steroid treatment adopted (dexamethasone yes vs no)
* Document any delays in the initiation of consolidation chemotherapy in LLA patients with IFI
* Document the outcome of patients with ALL with IFI

Study design The study is prospective and observational, multicenter, real-life study involving 26 centers afferent to the SEIFEM group. All Ph-neg ALL patients aged 18 years or older treated with intensive chemotherapy starting from 01.06.22 for the duration of 18 months (+12 months follow-up) will be enrolled. The diagnosis of IFI will be defined according to EORTC 2019 criteria. Clinical information will be collected in paper CRFs, compiled anonymously.

The incidence of IFI and pulmonary aspergillosis during induction chemotherapy will be related to the following variables:

* Age
* Sex
* Type of AF prophylaxis performed
* LLA risk classification according to ESMO 2016 criteria
* Dose of dexamethasone administered
* Duration of neutropenia
* Hematologic and molecular response

Inclusion criteria

* Patients with ALL B Ph-neg or T at onset
* Age > 18 yr at the time of the study
* Signature informed consent Exclusion criteria
* Patients with Ph-pos ALL
* Patients with relapsing ALL
* Patients with B/T lymphoblastic lymphoma Primary endpoint
* Incidence of IFI during the early stages of chemotherapy (from onset to TP2, i.e., week 16) in Ph-neg ALL patients.

Secondary endpoints

* Incidence of IFI in Ph-neg ALL patients during induction in relation to antifungal prophylaxis adopted
* Incidence of IFI in patients with Ph-neg ALL during induction in relation to age
* Incidence of IFI in Ph-neg ALL patients during induction in relation to duration of neutropenia
* Incidence of IFI in Ph-neg ALL patients in relation to type of steroid treatment adopted (dexamethasone yes vs no)
* Median time elapsed between actual start of consolidation chemotherapy versus schedule in Ph-neg ALL patients with IFI
* Patient mortality rate in Ph-neg ALL patients with IFI Study Duration All eligible patients will be enrolled from 01.03.2022 for a duration of 18 months. The follow-up time after enrollment will be 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with B Ph-neg or T ALL at onset
* Age > 18 yr at the time of the study
* Signature informed consent

Exclusion Criteria:

* Patients with Ph-pos ALL
* Patients with relapsing ALL
* Patients with B/T lymphoblastic lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by Ph-pos ALL
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-04-14 (Actual); Primary Completion 2024-03-12 (Actual); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of IFI during the early stages of chemotherapy (from onset to TP2, i.e., week 16) in Ph-neg ALL patients | 16 weeks
  Incidence of IFI during the early stages of chemotherapy (from onset to TP2, i.e., week 16) in Ph-neg ALL patients

SECONDARY OUTCOMES:
- Incidence of IFI in Ph-neg ALL patients during induction in relation to antifungal prophylaxis adopted | 16 weeks
  - Incidence of IFI in Ph-neg ALL patients during induction in relation to antifungal prophylaxis adopted
- Incidence of IFI in patients with Ph-neg ALL during induction in relation to age | 16 weeks
  - Incidence of IFI in patients with Ph-neg ALL during induction in relation to age
- Incidence of IFI in Ph-neg ALL patients during induction in relation to duration of neutropenia | 16 weeks
  - Incidence of IFI in Ph-neg ALL patients during induction in relation to duration of neutropenia
- Incidence of IFI in Ph-neg ALL patients in relation to type of steroid treatment adopted (dexamethasone yes vs no) | 16 weeks
  - Incidence of IFI in Ph-neg ALL patients in relation to type of steroid treatment adopted (dexamethasone yes vs no)
- Median time elapsed between actual start of consolidation chemotherapy versus schedule in Ph-neg ALL patients with IFI | 16 weeks
  - Median time elapsed between actual start of consolidation chemotherapy versus schedule in Ph-neg ALL patients with IFI
Patient mortality rate in Ph-neg ALL patients with IFI | 16 weeks
  Patient mortality rate in Ph-neg ALL patients with IFI

CONTACTS AND LOCATIONS:
Overall Officials: chiara cattaneo, md, Principal Investigator — ASST Spedali Civili di Brescia
Locations (1):
- ASST degli Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2022-03-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT06392581/Prot_000.pdf